CLINICAL TRIAL: NCT01579578
Title: A Phase IIa Multi-centre Randomised Double-Blind Placebo-controlled Study to Assess the Efficacy, Safety and Pharmacokinetics of AZD8931 in Combination With Paclitaxel Versus Paclitaxel Alone in Patients With Metastatic, Gastric or Gastro-oesophageal Junction, Cancer Who Progress Following First Line Therapy and Are Ineligible for Treatment With Trastuzumab by HER2 Status (SAGE)
Brief Title: Assess the Efficacy of AZD8931 in Combination With Paclitaxel Versus Paclitaxel Alone in Patients With Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AstraZeneca sponsored trials of AZD8931 have been halted
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D0102C00006
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Metastatic, Gastric or Gastro-oesophageal Junction, Cancer
Keywords: Metastatic Gastric Cancer who progress following First Line Therapy and are Ineligible for Treatment with trastuzumab by HER2 Status
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — AZD 8931; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8931; Drug: Paclitaxel
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD8931 — 40 mg, oral dose twice daily
  Arms: 1
Drug: Placebo — Placebo, oral dose twice daily
  Arms: 2
Drug: Paclitaxel — IV once weekly for 3 weeks followed by a week off.

SUMMARY:
The purpose of the study is to assess the efficacy and safety and PK of AZD8931 plus paclitaxel versus paclitaxel alone in patients with metastatic, gastric or gastro-oesophageal junction, cancer.

DETAILED DESCRIPTION:
A Phase IIa Multi-centre Randomised Double-Blind Placebo-controlled Study to Assess the Efficacy, Safety and Pharmacokinetics of AZD8931 in Combination with Paclitaxel versus Paclitaxel alone in Patients with Metastatic, Gastric or Gastro-oesophageal Junction, Cancer who progress following First Line Therapy and are Ineligible for Treatment with trastuzumab by HER2 Status (SAGE)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older (20 years or older in Japan)
* Patients must have radiologically confirmed progression following 1st line fluoropyrimidine and platinum based treatment for metastatic gastric cancer (the date of progression and start of first line treatment to be captured on the database)
* Suitable for paclitaxel therapy.
* At least one lesion, not previously irradiated and not chosen for a mandatory fresh tumour biopsy during the study screening period, that can be accurately measured at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for accurate repeat assessment.
* Ineligible for trastuzumab treatment by local assessment. This should include IHC analysis to determine HER2 status with further testing by FISH/CISH when considered part of local practice. Eligible patients are defined as; HER2 IHC 0, HER2 IHC +1 and +2

Exclusion Criteria:

* Have received more than 1 prior chemotherapy regimen for metastatic gastric cancer. (chemotherapy as adjuvant treatment is permitted).
* Any prior taxane therapy (at any time from diagnosis of gastric cancer)
* Any prior therapy with an inhibitor of ErbB1 (EGFR) or ErbB2 (HER2) (eg, lapatinib)
* Resting ECG with measurable QTc(F) interval of greater than 480 msec at 2 or more time points within a 24 hour period (see section 6.4.9.1 )
* Unresolved toxicity grater than CTCAE grade 2 (except alopecia) from previous anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, M. D., Study Director — Scarborough General Hospital
Locations (15):
- Germany (2):
  - Research Site, Cologne
  - Research Site, Hamburg
- Japan (5):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kawasaki-shi
  - Research Site, Matsuyama
  - Research Site, Sapporo
- South Korea (3):
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Valencia
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

REFERENCES:
- See also: D0102C00006_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1625&filename=D0102C00006_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the early stopping of this study as a result of the AZD8931 program being stopped, the full planned enrolment was not carried out. This study was stopped after 39 were enrolled, 25 of whom were treated, which is less than the number planned in the protocol.
Pre-assignment Details: Due to the early stopping of this study as a result of the AZD8931 program being stopped, the full planned enrolment was not carried out. This study was stopped after 39 were enrolled, 25 of whom were treated, which is less than the number planned in the protocol.
Groups:
- AZD8931 40mg + Paclitaxel: AZD8931 40 mg bd (Twice daily) administered orally in combination with paclitaxel 80 mg/m2 administered intravenously [approximately 1 hour duration] on D1, 8 and 15 of each 28 day treatment cycle
- Placebo + Paclitaxel: AZD8931 matching placebo bd administered orally in combination with paclitaxel 80 mg/m2 administered intravenously [approximately 1 hour duration] on D1, 8 and 15 of each 28 day treatment cycle
Period: Overall Study
Arm/Group | AZD8931 40mg + Paclitaxel | Placebo + Paclitaxel
Started | 13 | 12
Ongoing | 3 | 0
Completed | 0 | 0
Not Completed | 13 | 12
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Eligibility criteria | 3 | 9
Not completed — Ongoing | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8931 40mg + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (8.71) [45 to 72] | 62.7 (13.60) [34 to 76] | 60.2 (11.34) [34 to 76]
Age, Customized [Number; unit: Participants] — Age Group
  Participants
    18 - < 50 years | 3 | 2 | 5
    50 - < 65 years | 7 | 4 | 11
    65 - < 75 years | 3 | 5 | 8
    >= 75 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnic Group Summary
  Participants
    Asian (Other Than Chinese or Japanese) | 8 | 7 | 15
    Chinese | 1 | 2 | 3
    Japanese | 4 | 3 | 7
HER2 Status: HER2/IHC (Local Assessment) [Number; unit: Participants] — HER2 Status (Local Labs): HER2/IHC (Local Assessment)
  Participants
    HER2 0 No staining/membrane staining <10% of cells | 8 | 6 | 14
    HER2 1+ Faint membrane staining ≥10% of cells | 3 | 5 | 8
    HER2 2+ Weak/moderate membrane staining ≥10% cells | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumour Size at 8 Weeks Were Analyzed for Comparing Relative Efficacy of AZD8931 Plus Paclitaxel With Paclitaxel Alone
Time Frame: Baseline and 8 weeks, accessed up to data cut off on 4 December 2012
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percentage change
Units Other Than Participants: change from baseline
Groups:
- AZD8931 + Paclitaxel: AZD8931 40 mg bd (Twice daily) administered orally in combination with paclitaxel 80 mg/m2 administered intravenously [approximately 1 hour duration] on D1, 8 and 15 of each 28 day treatment cycle
Arm/Group | AZD8931 + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 11 | 11
Number analyzed (change from baseline) | 8 | 9
percentage change | -7.7 (8.60) | -2.7 (8.64)
Statistical Analysis 1: Comparison: AZD8931 + Paclitaxel vs Placebo + Paclitaxel; 60 patients had been considered to detect a -20% difference in the estimated average percentage change in tumour size at 8 weeks for AZD8931 plus paclitaxel compared to paclitaxel alone at a one-sided significance level of 10% with 90% power. This is based on a standard deviation of 30% for tumour data (on an absolute scale); Test type: Superiority or Other; p = 0.688, ANCOVA — two sided p value; ANCOVA model including covariates for baseline tumour size, for the time from the baseline scan to randomisation and with a term for HER2 status; Mean Difference (Final Values) = -5.00, 95% CI 2-sided [-30.81 to 20.81], Standard Error of Mean 12.23 — the difference in LS means is estimated

2. Secondary Outcome: Progression-free Survival (PFS) Were Analysed for Comparing Relative Efficacy of AZD8931 Plus Paclitaxel With Paclitaxel Alone
Description: Time from the date of randomization until the date of objective disease progression (as per RECIST1.1) or the date of death (by any cause in absence of progression).
Time Frame: Baseline and every 8 weeks, accessed up to data cut off on 4 December 2012
Measure: Median (Inter-Quartile Range); unit: months
Units Other Than Participants: events
Arm/Group | AZD8931 + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 13 | 12
Number analyzed (events) | 8 | 8
months | 3.7 [1.2 to 5.3] | 3.5 [1.7 to 5.1]

3. Secondary Outcome: The Objective Response Rate (ORR) Was Analysed for Investigating the Efficacy of AZD8931 Plus Paclitaxel With Paclitaxel Alone
Description: The number of subjects with at least one visit response of CR or PR. (Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive disease (PD), A ≥ 20% increase in the sum of diameters of target lesions and an absolute increase of ≥ 5mm; Stable disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Not Evaluable (NE), All target lesion measurements are missing or >1/3 target lesion measurements are missing and sum of diameters of non-missing target lesions does not qualify for PD; Not applicable (NA), No target lesions are recorded at baseline)
Time Frame: Baseline and 8 weeks, accessed up to data cut off on 4 December 2012
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | AZD8931 + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 13 | 12
Participants
  Total | 3 | 0
  Complete Response | 0 | 0
  Partial Response | 3 | 0

ADVERSE EVENTS:
Time Frame: AEs will be collected from time of signed informed consent throughout the treatment period and for 30 days after the last dose of AZD8931 /placebo
Arm/Group | AZD8931 40mg + Paclitaxel | Placebo + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 6/13 | 3/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 40mg + Paclitaxel (N=13) | Placebo + Paclitaxel (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 40mg + Paclitaxel (N=13) | Placebo + Paclitaxel (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 4 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 3 (9)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Accommodation disorder (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Scleral discolouration (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (13) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Asthenia (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 5 (5) | 4 (5)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (4)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (2)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (4)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 2 (4)
Weight decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (8) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (7)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Vulval oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (2)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days